CLINICAL TRIAL: NCT00506285
Title: Methylphenidate Transdermal System (MTS) in the Treatment of Adult ADHD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Shire (Industry)
Responsible Party: Principal Investigator, frederick reimherr, Associate Professor of Psychiatry, University of Utah
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20405; SPD485.420-Reimherr (Other Grant/Funding Number: Shire Pharma)
Record Dates: First submitted 2007-07-23; First posted 2007-07-25 (Estimated); Results first posted 2015-01-16 (Estimated); Last update posted 2015-01-16 (Estimated); Status verified 2015-01

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Attention Deficit Hyperactivity Disorder; ADHD; Adult; Methylphenidate Transdermal System; Daytrana
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): This arm was 4 weeks long. Subjects were treated using Methylphenidate Transdermal System. Patients were seen weekly, phone contact was made between visits and dosing could be adjusted as a result of the phone contact. MTS was initiated using a 12.5 cm patch. The dose was increased during the first 2 weeks based on treatment response and side effects to the largest tolerated dose/patch size. It was held steady the last 2 weeks.
  Interventions: Drug: Methylphenidate Transdermal System (MTS)
- B (Placebo Comparator): This arm was 4 weeks long. Placebo patch was initiated using a 12.5 cm patch and then increased to the largest tolerated patch size during the first 2 weeks and held steady the last two weeks. Subjects were seen weekly, phone contact was made between visits and dosing could be adjusted as a result of the phone visit.
  Interventions: Other: placebo patch

INTERVENTIONS:
Drug: Methylphenidate Transdermal System (MTS) — MTS is an advanced patch product that provides methylphenidate evenly mixed with the adhesive. This formulation allows good adhesion and a wide range of dose sizes. MTS patch sizes of 12.5, 18.75, 25 and 37.5cm2 are equivalent to nominal doses over a 9-hour wear time of 10, 15, 20 and 30mg of MPH.
  Other Names: Daytrana
  Arms: A
Other: placebo patch — This patch is designed to appear identical to the actual intervention patch
  Arms: B

SUMMARY:
This study will look at the effectiveness of Methylphenidate Transdermal System (MTS) in treating adult ADHD. MTS has received FDA approval for childhood ADHD but this is the first trial for adult ADHD. Subjects will experience two screening visits and one baseline visit. Those who meet admission criteria will enter the double-blind phase. This will involve two 4-week treatment periods one of which will involve the use of MTS and the other a placebo patch. Subjects who complete the double-blind phase will be allowed to enter a 180-day, open-label MTS phase designed to assess long-term effects.

DETAILED DESCRIPTION:
ADHD affects from 3 to 5% of children, persists into adolescence in 40 to 70% of these children and continues into adulthood in at least 50% of affected adolescents. Methylphenidate was the first medication shown to be effective in treatment for adults with ADHD and continues to be widely used. While the extended release formulations represent an improvement over the immediate release versions, significant problems remain for many patients. In particular, most have been designed with the goal of providing medication only during school hours and a short time period after school. In adults, there is a frequent need for much more extended duration of treatment. MTS is a new form of methylphenidate that provides medication in a transdermal patch delivery system. It has a very even, slowly ascending pharmacokinetic profile. MTS's very stable slowly increasing blood level should overcome the problems noted above with a delivery system that is more convenient for many patients. It is currently approved for treatment of childhood ADHD, with effectiveness and safety profiles similar to other forms of methylphenidate. This study will be the first to evaluate the effectiveness and safety of MTS in adult ADHD.

This is a double-blind, placebo-controlled, randomized, crossover trial comparing MTS with placebo patch. The double-blind trial will be preceded by an enrollment period consisting of two screening visits followed as quickly as possible by a baseline visit. Patients who continue to meet admission criteria at baseline will be randomized into the first of two 4-week treatment periods. We will attempt to reach the highest tolerated dose size of MTS within 2 weeks and then observe the response over the last two weeks of each crossover phase. The double-blind period will be followed by a 180 day open-treatment, flexible-dose phase designed to assess long-term effects.

ELIGIBILITY:
Inclusion Criteria:

Adults meeting DSM-IV-Text Revision criteria for ADHD, the Utah Criteria for ADHD, and experiencing at least moderate impairment (a score of 4 or greater on the CGI-Severity Scale for ADHD at both Screening and Baseline visits) will be enrolled. Other criteria include:

1. Subjects ages 18 to 65, inclusive;
2. Female subjects are eligible to enter and participate in this study only if:

   1. She is of non-childbearing potential; has a male sexual partner who is surgically sterilized; is on implant of levonorgestrel, injectable progesterone, or an oral contraceptive; has an intrauterine device (IUD); or is sexually inactive with a male partner.
   2. Or agrees to use a double barrier method of contraception (any combination of physical and chemical methods) and has a negative urine pregnancy test at screening interview.
3. Subject must be in general good health as determined by medical history, ECG, and other analysis that, in the judgment of the study physician, would confirm the patient's good health.
4. Subjects must read and write at a level sufficient to provide written informed consent and complete study-related materials.

Exclusion Criteria:

* Subjects will not be eligible for inclusion in this study if any of the following criteria apply:

  1. Subjects with other current DSM-IV Axis I Disorders including Current or lifetime history of psychosis, current bipolar disorder type I, current Major Depressive Disorder, and Current Anxiety Disorder (unless in the opinion of clinic physician ADHD is the primary disorder and causes the disability seen in the patient);
  2. Subjects with any other DSM-IV Axis II diagnosis so severe that it would suggest non-responsiveness to pharmacotherapy for ADHD or noncompliance with the protocol;
  3. Subjects at risk for suicide or a risk to harm others;
  4. History of Substance Dependence according to DSM-IV criteria within 3 months of screening;
  5. Subjects currently abusing illegal drugs or alcohol are excluded from the study;
  6. Positive urine screen for drugs of abuse at screening for patients who have a significant history of substance use but still meet criteria 4 and 5. Patients not at risk for substance abuse will not be given a urine drug screen;
  7. Subjects in whom stimulants would represent a risk such as those with a history of stimulant abuse,
  8. History of uncontrolled hypertension or significant cardiovascular disease;
  9. Any known or suspected significant medical or psychiatric illnesses (e.g., hepatic or renal insufficiency, pulmonary (asthma, COPD, etc), gastrointestinal, endocrine, neurological or metabolic disturbances that, in the judgment of the investigator, may impair interpretation of study results or constitute a significant safety concern in the context of the clinical trial;
  10. Medications, including health food supplements judged by the investigator to be likely to have central nervous system activity (for example, St John's Wort, gingko leaf, and melatonin), are not permitted during the study. If the subject is taking the medication prior to study entry, there must be a 7 day washout period prior to Visit 2. We will ask for an honest report of all medications consumed between visits. In the event a medication with psychoactive properties is consumed, the patient will be counseled regarding the use of prohibited medications;
  11. Use of any medication not considered acceptable by the clinical investigator or the medical monitor during the 7-day period before the start of the study (Day 1);
  12. Subjects with high BMI (>38) and those with high adipose tissue concentrations in the hip as judged by the clinician.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2007-06; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frederick W. Reimherr, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah School of Medicine, Department of Psychiatry, Mood Disorders Clinic, Salt Lake City, Utah, United States

REFERENCES:
- [Background] Olsen JL, Reimherr FW, Marchant BK, Wender PH, Robison RJ. The effect of personality disorder symptoms on response to treatment with methylphenidate transdermal system in adults with attention-deficit/hyperactivity disorder. Prim Care Companion CNS Disord. 2012;14(5):PCC.12m01344. doi: 10.4088/PCC.12m01344. Epub 2012 Oct 11. PMID 23469326
- [Result] Reimherr FW, Marchant BK, Olsen JL, Wender PH, Robison RJ. Oppositional defiant disorder in adults with ADHD. J Atten Disord. 2013 Feb;17(2):102-13. doi: 10.1177/1087054711425774. Epub 2011 Nov 18. PMID 22100691
- [Derived] Gift TE, Reimherr FW, Marchant BK, Steans TA, Wender PH. Personality Disorder in Adult Attention-Deficit/Hyperactivity Disorder: Attrition and Change During Long-term Treatment. J Nerv Ment Dis. 2016 May;204(5):355-63. doi: 10.1097/NMD.0000000000000470. PMID 27082828

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects (n=92) were recruited from 4-16-2007 through 10-24-2008. They were seen at the Psychiatry Research Clinic at the University of Utah School of Medicine.
Pre-assignment Details: There were 3 screening visits. Subjects met DSM-IV &/or Utah criteria for adult ADHD, experiencing at least moderate impairment. Most DSM-IV axis-I disorders were excluded. Of 92 subjects enrolled, 65 were randomized and produced double-blind data. The assessment procedure was more extensive than normal, leading to a high dropout rate.
Groups:
- A) MTS Arm Was 1st and PBO Arm Was 2nd: MTS was initiated using a 12.5cm2 patch then increased to the highest possible tolerated dose within two weeks and held at that level for the final two weeks of the first 4-week arm. In the second double-blind arm subjects were started using a 12.5cm2 placebo patch, which was increased to the highest tolerated dose within two weeks and held at that level for the final two weeks of the second 4-week arm.
- B) PBO Arm Was 1st and MTS Arm Was 2nd: Placebo was initiated using a 12.5cm2 patch then increased to the highest possible tolerated dose within two weeks and held at that level for the final two weeks of the first 4-week arm. In the second double-blind arm subjects were started using a 12.5cm2 MTS patch, which was increased to the highest tolerated dose within two weeks and held at that level for the final two weeks of the second 4-week arm.
Period: 3 Week Screening Phase
Arm/Group | A) MTS Arm Was 1st and PBO Arm Was 2nd | B) PBO Arm Was 1st and MTS Arm Was 2nd
Started | 46 | 46
Completed | 29 | 36
Not Completed | 17 | 10
Not completed — Withdrawal by Subject | 17 | 10
Period: Double Blind Cross-Over Phase
Arm/Group | A) MTS Arm Was 1st and PBO Arm Was 2nd | B) PBO Arm Was 1st and MTS Arm Was 2nd
Started | 29 | 36
Received at Least 1 Dose MTS | 29 | 31
Completed | 20 | 31
Not Completed | 9 | 5
Not completed — Withdrawal by Subject | 4 | 3
Not completed — Lost to Follow-up | 5 | 2
Period: 6-month Open Label Phase
Arm/Group | A) MTS Arm Was 1st and PBO Arm Was 2nd | B) PBO Arm Was 1st and MTS Arm Was 2nd
Started | 20 | 31
Completed | 10 | 19
Not Completed | 10 | 12
Not completed — Lost to Follow-up | 1 | 7
Not completed — Withdrawal by Subject | 9 | 5

BASELINE CHARACTERISTICS:
Groups:
- a) Methylphenidate Transdermal System Was Taken First: Subjects took Methylphenidate Transdermal System in the first treatment arm and placebo patch in the second treatment arm
- B Placebo Patch Was Used First: Placebo patch was used in the first treatment arm and MTS in the second treatment arm.
- Total: Total of all reporting groups
Arm/Group | a) Methylphenidate Transdermal System Was Taken First | B Placebo Patch Was Used First | Total
Number analyzed (Participants) | 29 | 36 | 65
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 36 | 65
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.4 (9.5) | 40.4 (11.8) | 35.2 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 13 | 21
  Male | 21 | 23 | 44
Region of Enrollment [Number; unit: participants]
  United States | 29 | 36 | 65
Wender-Reimherr Adult Attention Deficit Disorder Scale [Mean (Standard Deviation); unit: units on a scale] — This is a investigator rated scale of ADHD symptoms. It assessed the 7 domains of the Utah Criteria using scores of 0 (none) to 4 (highly symptomatic). Total possible scores range from 0 (no symptoms) to 28 (worst possible score).
  units on a scale | 21.5 (4.2) | 21.3 (4.1) | 21.4 (4.2)

OUTCOME MEASURES:

1. Primary Outcome: Wender Reimherr Adult Attention Deficit Disorder Scale
Description: This scale measures the 7 domains of the Utah Criteria for Adult ADHD. Total scores run from 0 to 28. Normative samples average below 5. The worst possible score is 28.
Time Frame: Double-blind endpoints during MTS and placebo arms
Population: All subjects given active treatment "last observation carried forward" using a mixed models design.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Scores in MTS Arm: Average WRAADDS scores at end of active treatment (MTS) arm
- Scores in Placebo Arm: Average WRAADDS scores at end of placebo arm
Arm/Group | Scores in MTS Arm | Scores in Placebo Arm
Number analyzed (Participants) | 49 | 49
units on a scale | 11.0 (7.4) | 17.9 (6.6)
Statistical Analysis 1: Comparison: Scores in MTS Arm vs Scores in Placebo Arm; Test type: Non-Inferiority or Equivalence — F(1,47)=26.7, p=.001; p = .001, Mixed Models Analysis; F(1,47)=26.7, p=.001

2. Secondary Outcome: Conners' Adult ADHD Rating Scales (CAARS)
Description: Measures the DSM based ADHD criteria of Inattention and Hyperactivity/Impulsivity. There are 30 items scored 0-3 for a minimum score of 0 (no symptoms) and a maximum score of 90 worst possible symptoms.
Time Frame: Double-blind endpoints for MTS and placebo arms
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Scores in MTS Arm: Average CAARS score at end of active treatment
- Scores in Placebo Arm: Average CAARS score at end of placebo treatment
Arm/Group | Scores in MTS Arm | Scores in Placebo Arm
Number analyzed (Participants) | 49 | 49
units on a scale | 30.8 (19.1) | 49.5 (18.8)
Statistical Analysis 1: Comparison: Scores in MTS Arm vs Scores in Placebo Arm; Test type: Non-Inferiority or Equivalence — mixed models analysis; p = .001, Mixed Models Analysis — F(1,47)=24.8, p=.001

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during both double-blind treatment arms. Each arm was 4 weeks long. Subjects who did not complete the double-blind phase were included in the assessment.
Description: A list of likely AEs were assessed at each visit. In addition, the investigator recorded any additional concerns by the subjects.
Groups:
- MTS Arm: Adverse events and Serious AEs during active treatment (MTS) arm
- Placebo Arm: Adverse events and Serious AEs during placebo arm
Arm/Group | MTS Arm | Placebo Arm
Serious Adverse Events (participants affected / at risk) | 0/61 | 0/58
Other Adverse Events (participants affected / at risk) | 24/61 | 10/58
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MTS Arm (N=61) | Placebo Arm (N=58)
insomnia/sleep (General disorders) | 19 (19) | 4 (4)
dry eyes, nose, mouth (General disorders) | 8 (8) | 1 (1)
headache (General disorders) | 8 (8) | 4 (4)
anxiety (General disorders) | 7 (7) | 1 (1)
decreased appetite (Gastrointestinal disorders) | 7 (7) | 2 (2)
anger/irritability (Psychiatric disorders) | 7 (7) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No